CLINICAL TRIAL: NCT02537405
Title: Randomized, Non-blinded, Two-way Crossover Study to Establish the Bioequivalence Between a Rivaroxaban Tablet 10 mg and a Rivaroxaban Granule 10 mg in Japanese Healthy Adult Male Subjects
Brief Title: Bioequivalence Study of Rivaroxaban in Japanese Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17018
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Embolism, Atrial Fibrillation and Venous Thrombosis
MeSH Terms: conditions — Embolism; Atrial Fibrillation; Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAY59-7939 granule (Experimental)
  Interventions: Drug: Rivaroxaban (BAY 59-7939)
- BAY59-7939 tablet (Active Comparator)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY 59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (BAY 59-7939) — Rivaroxaban granule 10mg for one day
  Arms: BAY59-7939 granule
Drug: Rivaroxaban (Xarelto, BAY 59-7939) — Rivaroxaban tablet 10mg for one day
  Arms: BAY59-7939 tablet

SUMMARY:
The objectives of this study are to establish the bioequivalence between rivaroxaban tablet 10mg and rivaroxaban granule formulation 10mg, and to assess the safety and tolerability of rivaroxaban 10mg in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male subjects
* 20 to 40 years of age
* 17.6 to 26.4 kg / m² of body mass index (BMI)

Exclusion Criteria:

* Subject with incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Subject with a history of relevant diseases of vital organs, of the central nervous system or other organs, eg instable coronary heart disease, heart failure, liver failure, kidney failure, hypotension, or history of stroke or myocardial infarction
* Subject with known coagulation disorders (eg von Willebrand's disease, hemophilia)
* Subject with known disorders with increased bleeding risk (eg periodontosis, hemorrhoids, acute gastritis, peptic ulcer)
* Subject with known sensitivity to common causes of bleeding (eg nasal)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed drug concentration in measured matrix after single dose administration) | Multiple time point up to 3 day
AUC(0-tlast) (AUC from time 0 to the last data point > LLOQ (lower limit of quantitation)) | Multiple time point up to 3 day

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kumamoto, Kumamoto, Japan